CLINICAL TRIAL: NCT05560451
Title: Telehealth-delivered Peer Support to Improve Quality of Life Among Veterans With Multimorbidity
Acronym: VetASSIST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 21-100
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Multimorbidity
Keywords: Peer health coaching; Health-related quality of life; Veterans; Multimorbidity; Self-management; Social support; Multiple chronic conditions; Telemedicine
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Intervention Model Description: Hybrid type 1 trial with 294 Veterans with multimorbidity. Participants will be randomized to one of two groups -- the control or intervention group -- in parallel for the duration of the study.
Who Masked: Outcomes Assessor
Masking Description: Concealment will be used to prevent the study staff from obtaining information on the sequence of assignment. Because of the nature of the intervention, we are unable to blind participants and staff to treatment assignment. Staff who complete outcomes assessment are masked to study assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peer health coach intervention (Experimental): Participants will receive 20 virtual visits with a trained Veteran peer health coach over 12 months. Coaches will provide participants with brief health education, assist with goal setting and problem solving, enhance social support, and link participants to VA and community resources.
  Interventions: Behavioral: Peer health coach intervention
- Control group/no intervention (No Intervention): Participants will continue to receive their regular, usual primary care.

INTERVENTIONS:
Behavioral: Peer health coach intervention — Eligible participants will be randomly assigned to receive a telehealth delivered peer health coach intervention to promote health outcomes and behavior change among Veterans with multimorbidty.
  Other Names: VetASSIST
  Arms: Peer health coach intervention

SUMMARY:
The VetASSIST study is a randomized clinical trial testing whether receiving virtual health coaching from Veteran peers improves the physical and mental health-related quality of life of Veterans with multiple chronic health conditions and complex healthcare needs. VetASSIST will test the efficacy of an intervention that matches Veteran patients with multimorbidty with Veteran health coaches who will provide education, resources, guidance and support to help them manage their physical and mental health over the course of a year.

DETAILED DESCRIPTION:
The study objective is to evaluate the effectiveness of a virtual, Veteran peer-led self-management support program (VetASSIST) to improve health related quality of life (HRQoL) for Veterans with multimorbidity compared to usual care. The investigators will conduct a type 1 hybrid effectiveness-implementation randomized controlled trial of the intervention among VA Puget Sound patients with multimorbidity. Trained peer health coaches will virtually meet one-on-one with patients to assist in daily self-management by providing information; identifying patients' values and preferences; helping them set goals in alignment with their values and preferences and problem-solve barriers to those goals; modeling skills for effective management; providing social support; linking them to clinical care and community resources; and addressing self-management barriers. Veterans with multimorbidity will be randomized to receive the peer health coaching intervention or usual care. Outcomes will be assessed remotely at baseline and 12 months.

Specific aims are: 1) Test the effect of VetASSIST, compared to usual care, on the primary outcome of baseline to 12-month change in physical HRQoL, and secondary outcomes of mental HRQoL and health care utilization; 2a) Describe differences between VetASSIST and usual care on baseline to 12-month changes in intermediate outcomes reflecting the functions of peer support and intervention targets (self-efficacy, patient activation, health behaviors, social support, perceived access to care, patient-provider communication, and shared decision-making); 2b) Examine whether intermediate outcomes mediate intervention-associated differences in HRQoL; 3) Evaluate feasibility of translating VetASSIST into practice, including evaluation of per patient intervention costs and barriers and facilitators to implementation.

ELIGIBILITY:
Inclusion Criteria:

* Veteran patient receiving primary care from VA Puget Sound
* Complex multimorbidity (>=3 chronic conditions in >=3 body systems based on AHRQ Chronic Condition Index)
* Meets >=2 criterion from NICE multimorbidity guidelines: 1) have a chronic physical and mental health condition (via ICD-10 codes in CDW and the CCI); 2) frailty (determined by the JEN Frailty Index available in VA data, confirmed via self-reported PRISMA-7 during the eligibility screening; 3) frequent emergency care (>=1 VA emergency department visit in past year via CDW); 4) polypharmacy (>=10 prescribed medications via CDW), or 5) significant treatment burden (score >22 on the self-reported Multimorbidity Treatment Burden Questionnaire at study screening).
* Inclusion criteria assessed via the phone screen includes frailty; treatment burden; and willingness to use a either a phone or an Internet-connected device with a web camera and an email address and/or ability to receive text messages to ensure receipt of VVC visit links.
* Agree to participate in the health coaching sessions and surveys if assigned to intervention group

Exclusion Criteria:

* Not fluent in English
* Severe hearing loss
* No phone access and/or missing phone number
* Missing address
* Diagnosis of dementia or severe cognitive impairment within last year
* Diagnosis of end stage renal disease or on dialysis within last year
* Receipt of palliative or hospice care in the past year
* Receipt of nursing home care in past year (Stop codes: 650, 651,119,121)
* Currently living in a nursing home, skilled nursing facility, rehabilitation facility, or long-term care facility
* Behavior flags in EHR
* Active treatment for non-melanoma skin cancer diagnosis
* Diagnosis of substance use dependence/abuse disorder in last year (excluding tobacco)
* Diagnosis of psychotic disorder in last year
* Pregnant or planning to become pregnant in next 6 months
* Score of >8 (severe risk) on self-reported AUDIT-C questions on eligibility screen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in physical health related quality of life (HRQoL) | Baseline to 12-months
  12 Item Short Form Health Survey (SF-12) Physical Component Summary: Summary scores for general health, physical functioning, role-physical, and bodily pain. Scaling scores will be assessed using published standardized scoring system procedures for the SF-12 found at: www.researchgate.net/publication/242636950_SF-12_How_to_Score_the_SF-12_Physical_and_Mental_Health_Summary_Scales

SECONDARY OUTCOMES:
Change in mental health quality of life (HRQoL) | Baseline to 12-months
  12 Item Short Form Health Survey (SF-12) Mental Component Summary: Summary scores for vitality, mental health, social functioning, and role-emotional. Scaling scores will be assessed using published standardized scoring system procedures for the SF-12 found at: www.researchgate.net/publication/242636950_SF-12_How_to_Score_the_SF-12_Physical_and_Mental_Health_Summary_Scales
Health care utilization | Baseline to 12-months
  Measured by VA clinical and administrative data and self-report responses (non-VA care), including primary care, specialty care, inpatient admissions, emergency department visits. A higher number of visits indicates greater utilization.

OTHER OUTCOMES:
Self-efficacy | Baseline to 12-months
  Measured by the Self-Efficacy to Manage Chronic Disease Scale to assess perceived capability to perform actions required to manage chronic diseases. Confidence is measured on a 10-point scale ranging from (1) not at all confident to (10) totally confident. A higher score indicates higher self-efficacy/confidence.
Patient activation | Baseline to 12-months
  Measured by the Consumer Health Activation Index (CHAI) to assess ability to take preventive actions, manage symptoms, find and use medical care, and work with health care providers. Responses are measured as low activation vs. not low activation on a 4-point scale ranging from almost always true (1) to almost never true (4). A higher score indicates lower activation.
Social support | Baseline to 12-months
  Medical Outcomes Study (MOS) 8-Item Social Support Survey Instrument will measure emotional, instrumental, informational, and appraisal of social support. Social Support is scored using a 5-point response scale ranging from none of the time (1) to all of the time (5). A higher score for an individual scale or overall support index indicates greater support.
Loneliness | Baseline to 12-months
  Three-Item UCLA Loneliness Scale will measure subjective feelings of being lonely or isolated. Responses are measured using a 3-point response scale ranging from hardly ever (1) to often (3). A higher score indicates greater loneliness.
Access to care | Baseline to 12-months
  Consumer Assessment of Healthcare Providers and Systems (CAHPS) - access to care- will measure getting timely appointments, care, and information. Responses are measured using a 4-point response scale ranging from never (1) to always (4). A higher score indicates increased access to care.
Patient-provider communication | Baseline to 12-months
  Consumer Assessment of Healthcare Providers and Systems (CAHPS) - patient-provider communication- will measure communication with physician and health care team. Responses are measured using a 4-point response scale ranging from never (1) to always (4). A higher score indicates greater communication.
Shared decision-making | Baseline to 12-months
  CollaboRATE will measure explanation of health issues; elicitation and integration of patient preferences. Responses are measured using a 10-point response scale ranging from no effort was made (0) to every effort was made (9). A higher score indicates greater shared decision making.
Diet quality | Baseline to 12-months
  Starting the Conversation brief dietary assessment and intervention scale will measure diet quality. Responses are measured using a 3-point response scale. Items have a score range of 0, 1, 2. The total ranges from scores of 0 to 16. A higher score indicates a less healthful diet.
Medication adherence | Baseline to 12-months
  Voils Domains of Subjective Extent of Nonadherence (DOSE-Nonadherence) Reasons for Nonadherence measure will identify possible reasons for nonadherence to prescribed treatment. Medication adherence is scored using a 5-point response scale ranging from none of the time (1) to all of the time (5). Higher scores indicate greater nonadherence.
Tobacco use | Baseline to 12-months
  Behavioral Risk Factor Surveillance System (BRFSS) Questionnaire will measure tobacco use. Questions will assess current tobacco use and frequency of use. Current tobacco use includes individuals who report having smoked at least 100 cigarettes in their entire life and who report smoking cigarettes now (every day or some days).
Alcohol use | Baseline to 12-months
  AUDIT Alcohol Consumption questionnaire (AUDIT-C) will measure alcohol use. A total of 5+ indicates increased or higher risk drinking. An overall total score of 5 or above is AUDIT-C positive.
Sleep impairment/disturbance | Baseline to 12-months
  PROMIS Sleep Related Impairment and Sleep Disturbance survey will measure sleep disturbance related impairment. Responses are measured on a 5-point scale ranging from not at all (1) to very much (5). A higher score indicates greater sleep disturbance.
Physical activity | Baseline to 12-months
  International Physical Activity Questionnaire (IPAQ) Short form assessment will measure physical activity. We will examine total physical activity in minutes per week, totaling all time from walking, moderate, and vigorous activity in the past 7 days. We will also examine physical activity dichotomously, identifying those meeting recommendations of at least 150 minutes total physical activity per week. We will use standard data cleaning procedures outlined by IPAQ developers, available at www.ipaq.ki.se.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen E. Gray, PhD MS BS, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA; Katherine D Hoerster, PhD MPH BA, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gray KE, Williams JL, Rivera-Remines A, Fennell T, Rao M, Rogers T, Taylor L, Nelson KM, Hoerster KD. Protocol for VetASSIST: A randomized controlled trial to evaluate virtual peer health coaching for veterans with multimorbidity. Contemp Clin Trials. 2025 Oct;157:108045. doi: 10.1016/j.cct.2025.108045. Epub 2025 Aug 14. PMID 40818733

DOCUMENTS (1):
  • Informed Consent Form (2025-08-07): https://cdn.clinicaltrials.gov/large-docs/51/NCT05560451/ICF_000.pdf